CLINICAL TRIAL: NCT00931814
Title: Effects of Exercise on Depression Symptoms, Physical Function, and Quality of Life in Community-Dwelling Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Ying-Tai Wu, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9461701114
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Healthy Elderly
Keywords: Depression; physical function; Quality of life
MeSH Terms: conditions — Depression | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exercise (Other)
  Interventions: Other: exercise training

INTERVENTIONS:
Other: exercise training — A progressive and structured, small-group exercise training 3 times a week, 30-40 min a session at intensity of 12-14 in rate of perceived exertion (RPE) for 8 weeks
  Other Names: exercise

SUMMARY:
The purpose of this study was to investigate the effects of 8-week exercise training on depression symptoms, physical functions, and quality of life in the community-dwelling elderly.

ELIGIBILITY:
Inclusion Criteria:

* elderly subjects living in the community aged 65 years or older, sedentary lifestyle

Exclusion Criteria:

* cancer, major neuromuscular disease, respiratory or cardiovascular disease which might affect exercise
* post myocardial infarction or major surgery in the previous year
* psychological disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-12; Primary Completion 2006-05 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Taiwanese Geriatric Depression Scale (TGDS), Mini-Mental State Examination (MMSE), Groningen Activity Restriction Scale (GARS) | 8 weeks

SECONDARY OUTCOMES:
Short-form 36 (SF-36) | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan